CLINICAL TRIAL: NCT00241930
Title: SPNS Buprenorphine and Integrated HIV Care Evaluation and Support Center: Integration of Buprenorphine and HIV Treatment Using the OASIS Model
Brief Title: Integrating Buprenorphine Into HIV Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organization to Achieve Solutions in Substance Abuse (OASIS) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H97HA03792; 1 H97HA03792-01-00
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-08

CONDITIONS: Opiate Dependence; HIV Infections
Keywords: Heroin; HIV; buprenorphine; integration; drug treatment
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections

INTERVENTIONS:
Behavioral: Integrating drug treatment into HIV services

SUMMARY:
We hypothesize that integrating drug treatment into HIV treatment will improve HIV outcomes as well as drug treatment outcomes in heroin users. This study will test this hypothesis by randomizing patients to two groups. The first group will receive HIV treatment and buprenorphine treatment contemporaneously at their HIV clinic. The second group will receive HIV treatment at their HIV clinic, and go to another facility to receive buprenorphine treatment services.

We will look at HIV outcomes such as CD4 counts, HIV viral loads, and attendance at appointments and drug treatment outcomes such as receipt of buprenorphine and urine toxicology testing.

DETAILED DESCRIPTION:
This study will test the hypothesis that integrating buprenorphine within the context of primary care HIV treatment will improve outcomes for HIV-infected heroin users vs providing buprenorphine services at a separate, off-site facility. As a means of engagement, we will offer the OASIS education group each week at each facility. For those randomized to integrated care, subjects will attend one education session weekly at the time of their HIV clinic. During these sessions, subjects will receive contemporaneous HIV clinic appointments (monthly), case management (monthly), drug counseling (twice monthly), and buprenorphine (which will be dispensed weekly.) For those randomized to separate care, subjects will attend HIV clinic appointments monthly, and will attend weekly education sessions at the OASIS facility. During these sessions, subjects will receive weekly buprenorphine, twice monthly drug counseling, and monthly case management.

We will measure outcomes by reporting attendance, CD4 counts, HIV viral loads, urine toxicology testing on at least a quarterly basis. We will also measure patient satisfaction, knowledge, quality of life, and a number of other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ as verified by lab report
* DSM-IV diagnosis of opioid dependence
* Speaks/understands English
* Age 18 years or older

Exclusion Criteria:

* LFT's (transaminase) >5x ULN
* DSV-IV criteria for benzodiazepine abuse or dependence within the last month
* DSM-IV criteria for alcohol dependence within the past 6 months
* Actively suicidal
* Methadone dose exceeds level allowing safe transition to buprenorphine
* Pregnant women and women trying to become pregnant
* Unable to provide informed consent
* Clinical judgement that patient is inappropriate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2009-02

PRIMARY OUTCOMES:
1.Impact of integrated care vs nonintegrated care on:
a. Substance use and high-risk transmission behaviors
b. Medical engagement and outcomes
c. Psychosocial indices, such as criminal justice, employment, housing, and education

SECONDARY OUTCOMES:
1. Acceptability of HIV treatment-based buprenorphine therapy
2. Health services utilization

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Sylvestre, MD, Principal Investigator — Organization to Achieve Solutions in Substance Abuse (OASIS); Ruth Finkelstein, ScD, Study Director — New York Academy of Medicine
Locations (3):
- United States (3):
  - Alameda County Medical Center HIV Clinic, Oakland, California
  - OASIS, Oakland, California
  - Fairmont Hospital HIV Clinic, San Leandro, California